CLINICAL TRIAL: NCT06929936
Title: Phase II Clinical Trial of Trilaciclib in Combination With Docetaxel for Second-Line and Beyond Treatment of Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Trilaciclib in Combination With Docetaxel for Second-Line and Beyond Treatment of Locally Advanced or Metastatic NSCLC
Acronym: PROTECT-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROTECT-1
Record Dates: First submitted 2025-03-23; First posted 2025-04-16 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Cancer; Myelosuppression
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trilaciclib combined with Docetaxel (Experimental): Trilaciclib combined with Docetaxel
  Interventions: Drug: Trilaciclib combined with Docetaxel

INTERVENTIONS:
Drug: Trilaciclib combined with Docetaxel — Trilaciclib: 240 mg/m2 as a 30-min iv. infusion, completed ≤4h prior to chemotherapy.
  Docetaxel: 75mg/m2, iv. infusion for 1 hour on days 1 of each 21-day cycle, totaling 4 cycles of medication.

SUMMARY:
This study is a prospective, single arm phase II study aimed at patients with locally advanced or metastatic non-small cell lung cancer undergoing second-line or beyond treatment. The aim is to evaluate the bone marrow protective effect of trilaciclib before docetaxel chemotherapy for locally advanced or metastatic NSCLC.

DETAILED DESCRIPTION:
After obtaining informed consent from patients diagnosed with locally advanced or metastatic NSCLC through pathology, 33 eligible subjects who met the inclusion criteria were selected to receive the treatment regimen of trilaciclib before docetaxel chemotherapy, with a treatment period of 4 cycles.

Record the dynamic changes of whole blood cell count; Hematological toxicity, including febrile neutropenia and associated infections; Transfusion of blood products and supplementation of hematopoietic raw materials. Perform tumor imaging evaluation according to RECIST 1.1. Baseline imaging examination shall be conducted within 21 days prior to the first administration, and tumor imaging evaluation shall be conducted every 6 weeks (± 7 days) from the first study drug administration, or the frequency of imaging evaluation may be increased when there are clinical indications. The imaging examination time should follow the calendar day and should not be adjusted due to treatment delay or termination. Subjects who terminate the study drug treatment due to intolerable toxicity or other non disease progression reasons should continue to receive tumor evaluation follow-up until disease progression, withdrawal from the study, or death (whichever occurs earliest)

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be included in this study:

1. Age ≥ 18 years old, regardless of gender;
2. Patients with stage IV NSCLC who have failed at least one line of standard treatment regimen:

   A. Patients with negative driver genes must have received first line standard treatment (chemotherapy combined with immunotherapy).

   B. Patients with positive driver genes must have received at least one line chemotherapy after standard targeted therapy has failed.

   C. Definition of driver genes: EGFR (including 19del, L858R, S768I, L861Q, and/or G719X), BRAF V600E, NTRK, MET14 exon skipping mutation, RET, ROS1, etc.
3. At least one measurable lesion that meets the RECIST 1.1 criteria exists;
4. The laboratory test results meet the following criteria:

   Hemoglobin ≥ 100 g/L (female), 110g/L (male) ,Neutrophil count ≥ 2×109/L Platelet count ≥ 100×109/L; Creatinine ≤15mg/L or creatinine clearance rate (CrCl) ≥ 60mL/min (Cockcroft Gault formula); Total bilirubin ≤ 1.5xupper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3×ULN or ≤ 5×ULN (for patients with liver metastases); Albumin ≥ 30 g/L;
5. ECOG PS score 0-2;
6. Expected survival time ≥ 3 months;
7. Women: All women with potential fertility must have a negative serum pregnancy test result during the screening period, and must take reliable contraceptive measures from signing the informed consent form until 3 months after the last dose;
8. Understand and sign the informed consent form.

Exclusion Criteria:

1. Previously received treatment with docetaxel;
2. Diagnosed with malignant diseases other than NSCLC within 5 years prior to the first administration (excluding curative basal cell carcinoma, squamous cell carcinoma, and/or excised carcinoma in situ);
3. Uncontrolled ischemic heart disease or clinically significant congestive heart failure (NYHA class III or IV);
4. Stroke or cardiovascular events within the first 6 months of enrollment;
5. When screening, if the QTcF interval is greater than 480 milliseconds, for patients implanted with ventricular pacemakers, QTcF>500msec；
6. Human immunodeficiency virus (HIV) infected individuals (HIV 1/2 antibody positive), known syphilis infected individuals;
7. Previously received hematopoietic stem cell or bone marrow transplantation;
8. Allergies to research drugs or their components;
9. The researchers believe that it is not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade ≥ 3 neutropenia during chemotherapy treatment | Time from date of first dose of trilaciclib and docetaxel through 30 days following the last dose of trilaciclib and docetaxel

SECONDARY OUTCOMES:
Incidence rate of grade 3 or 4 thrombocytopenia | Time from date of first dose of trilaciclib and docetaxel through 30 days following the last dose of trilaciclib and docetaxel
Incidence rate of grade 3 or 4 anemia during chemotherapy treatment | Time from date of first dose of trilaciclib and docetaxel through 30 days following the last dose of trilaciclib and docetaxel
Incidence rate of febrile neutropenia | Time from date of first dose of trilaciclib and docetaxel through 30 days following the last dose of trilaciclib and docetaxel
Usage rate of symptomatic treatments for myelosuppression | Time from date of first dose of trilaciclib and docetaxel through 30 days following the last dose of trilaciclib and docetaxel
  such as granulocyte colony-stimulating factor (G-CSF) (not for prevention), thrombopoietin (TPO), interleukin-11 (IL-11), erythropoiesis-stimulating agents (ESA), iron supplements, etc
Objective response rate | 12 months after the last subject participating in
Disease control rate | 12 months after the last subject participating in
Duration of response | 12 months after the last subject participating in
Progression-free survival | 12 months after the last subject participating in
Overall survival | From the date of randomization to the date of death for patients who died in the study due to any cause, or to the last contact date known to be alive for those who survived as of the data cutoff date, assessed up to 30 months.
Incidence rate of adverse events | Time from date of first dose of trilaciclib and docetaxel through 90 days following the last dose of trilaciclib and docetaxel

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes